CLINICAL TRIAL: NCT01002248
Title: A Phase III Randomized Study to Assess the Efficacy and Safety of Perifosine Added to the Combination of Bortezomib and Dexamethasone in Multiple Myeloma Patients
Brief Title: Assessment of Efficacy and Safety of Perifosine, Bortezomib and Dexamethasone in Multiple Myeloma Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Perifosine 339
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2013-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed multiple myeloma; Refractory multiple myeloma; Relapsed refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — perifosine; Bortezomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perifosine added to combination (Experimental): Perifosine added to the combination of Bortezomib and Dexamethasone. Perifosine is is supplied as a film-coated tablet containing 50 mg of active ingredient. Perifosine will be administered orally on an outpatient basis throughout the study. Daily administration will be one 50 mg tablet.
  The first dose of perifosine should be taken on the same day that bortezomib and dexamethasone are administered (Cycle 1 Day 1).
  Interventions: Drug: Perifosine; Drug: Bortezomib; Drug: Dexamethasone
- Perifosine Placebo added to combination (Placebo Comparator): Perifosine placebo added to the combination of Bortezomib and Dexamethasone. The placebo for perifosine is provided in 256 mg white to off-white, round, biconvex film-coated tablets to permit a blinded trial with perifosine 50 mg film coated tablets. Placebo will be administered orally on an outpatient basis throughout the study. Daily administration will be one perifosine placebo tablet. The first dose of placebo should be taken on the same day that bortezomib and dexamethasone are administered (Cycle 1 Day 1).
  Interventions: Drug: Perifosine Placebo; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Perifosine — Perifosine will be dosed as one 50 mg pill every day of each cycle.
  Other Names: D-21266; KRX-0401
  Arms: Perifosine added to combination
Drug: Perifosine Placebo — Perifosine placebo will be dosed as one 50 mg pill every day of each cycle.
  Arms: Perifosine Placebo added to combination
Drug: Bortezomib — Bortezomib will be dosed at 1.3 mg/m2 on Days 1, 4, 8, and 11 every 21 days.
Drug: Dexamethasone — Dexamethasone will be administered orally at 20 mg on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle.

SUMMARY:
This is a randomized Phase III study to evaluate the efficacy and safety of perifosine when added to the combination of bortezomib and dexamethasone in multiple myeloma patients who have relapsed on a prior bortezomib treatment regimen.

DETAILED DESCRIPTION:
A pre-planned interim analysis is expected to take place in Q1 of 2013.

ELIGIBILITY:
Inclusion Criteria:

* Patient was previously diagnosed with multiple myeloma based on standard diagnostic criteria.
* Patients must have relapsed (progressed > 60 days) after their last dose of bortezomib-based therapy. In addition, patients may be relapsed or refractory to other non-bortezomib-based therapies.
* Patient has received at least 1 but not more than 4 prior anti-myeloma regimens and has progressive disease after the most recent treatment regimen.
* Patients must have adequate organ and marrow function.

Exclusion Criteria:

* Patients must not be refractory to any bortezomib-containing regimen.
* History of allergic reactions or intolerance attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine), bortezomib or dexamethasone or any of their components.
* Prior treatment with perifosine or an investigational proteasome inhibitor.
* Chemotherapy or other therapy experimental or proven that is or may be active against myeloma within two weeks (14 days) prior to Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determine the PFS (progression free survival) in patients with multiple myeloma, treated with perifosine, bortezomib and dexamethasone compared to patients treated with placebo, bortezomib and dexamethasone | 6 - 24 months
  Progression-free survival will be defined as the time between randomization and the date of progression that occurred during the Core Phase.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months
  OS is defined as time from randomization to death from any cause during the Core Phase of the study.
Overall response rate (ORR) | 6 - 24 months
  The ORR for each treatment arm will be estimated as the proportion of responders, defined as a patient whose best overall response is PR or better during the treatment period, using criteria prospectively established.
Adverse Events | Up to 24 months
  Each AE and SAE term submitted will be mapped to a preferred term (PT) using the MedDRA dictionary. The investigator will classify the severity of AEs using the NCI CTCAE v3.0 and will assess the relationship of each event to each study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (72):
- United States (38):
  - La Verne, California
  - San Francisco, California
  - San Pablo, California
  - Aurora, Colorado
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Longmont, Colorado
  - Parker, Colorado
  - Pueblo, Colorado
  - Thornton, Colorado
  - Niles, Illinois
  - Winfield, Illinois
  - Baltimore, Maryland
  - Columbia, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Morristown, New Jersey
  - Great Neck, New York
  - Fargo, North Dakota
  - Portland, Oregon
  - Tualatin, Oregon
  - Kingsport, Tennessee
  - Bedford, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Kerrville, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Ogden, Utah
  - Christiansburg, Virginia
  - Roanoke, Virginia
  - Salem, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Vancouver, Washington
  - Milwaukee, Wisconsin
- Canada (3):
  - Winnipeg, Manitoba
  - Montreal, Quebec
  - Québec, Quebec
- Czechia (2):
  - Brno, Czech Republic
  - Prague, Czech Republic
- Ireland (7):
  - Keryx / AOI Pharmaceuticals Investigative Site, Dublin
  - Dublin
  - Galway
  - Limerick
  - Sligo
  - Tullamore
  - Waterford
- Israel (10):
  - Afula
  - Ashkelon
  - Beersheba
  - Haifa
  - Jerusalem
  - Nahariya
  - Petah Tikva
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Samara
- Košice, Slovak Republic, Slovakia
- Seoul, South Korea
- Spain (7):
  - Badalona
  - Barcelona
  - Madrid
  - Pamplona
  - San Cristóbal de La Laguna
  - Valencia
  - Zaragoza

REFERENCES:
- [Result] Richardson PG, Nagler A, Ben-Yehuda D, Badros A, Hari P, Hajek R, Spicka I, Kaya H, Le Blanc R, Yoon SS, Kim K, Martinez-Lopez J, Mittelman M, Shpilberg O, Tothova E, Laubach JP, Ghobria IM, Leiba M, Gatt ME, Sportelli P, Chen M, Anderson KC. Randomized Placebo-Controlled Phase III Study Of Perifosine Combined With Bortezomib and Dexamethasone In Relapsed, Refractory Multiple Myeloma Patients Previously Treated With Bortezomib. Blood 2013 ASH Meeting Proceedings;122:abstract 3189